CLINICAL TRIAL: NCT00339131
Title: Phase 1 Study Evaluating the Safety, Distribution, Metabolism, and Radiation Dosimetry of ULTRATRACE Iobenguane I 131 in Patients With Malignant Pheochromocytoma/Paraganglioma or Metastatic Carcinoid
Brief Title: ULTRATRACE Iobenguane I 131 in Patients With Malignant Pheochromocytoma, Paraganglioma, or Metastatic Carcinoid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIP-IB11
Record Dates: First submitted 2006-06-17; First posted 2006-06-20 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Pheochromocytoma; Paraganglioma; Carcinoid
Keywords: radiopharmaceutical; radiation dosimetry; iodine; MIBG; iobenguane; Ultratrace; neuroendocrine tumors
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Carcinoid Tumor; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ultratrace iobenguane I 131

SUMMARY:
The purpose of this study is to test the safety of a drug called Ultratrace iobenguane I 131 that has radioactivity, to measure how long it takes for the drug to be absorbed and passed out of the body, and to measure how much radioactivity is absorbed into different tissues of the body.

DETAILED DESCRIPTION:
Iobenguane, which is also known as MIBG, has been used in many patients who have types of cancers caused by what are known as neuroendocrine tumors, such as pheochromocytoma, paraganglioma, and carcinoid. Iobenguane is absorbed by neuroendocrine tumor cells. The radioactive portion of the study drug, Ultratrace iobenguane, is a form of iodine called I 131. The I 131 is absorbed into the tumor with the iobenguane, and the radioactivity should kill the tumors. The type of iobenguane being studied is called Ultratrace because of the new way in which this form of iobenguane is made. This study is the first time in which Ultratrace iobenguane will be given to patients. The purpose of the study is to give a low dose of iobenguane just to find out if the drug is safe, to measure how long it takes the drug to be absorbed and passed out of the body, and to see how much radioactivity is absorbed by different types of tissues of the body.

ELIGIBILITY:
Inclusion Criteria:

Patients will enter one of two study arms depending on their type of neuroendocrine tumor.

Arm P patients must:

* Have a biochemical or histopathological diagnosis of either adrenal pheochromocytoma or extra-adrenal paraganglioma (biochemical diagnosis includes plasma-free metanephrines and 24-hour urine test for catecholamines/metanephrines)
* Disease is metastatic or has recurred following surgery
* Have a CT scan performed (for later measurement of disease volume by the core lab) within 90 days of the administration of study drug without any interventions between CT and iobenguane I 131 imaging.

Arm C patients must:

* Have a histopathological diagnosis of carcinoid, or by plasma chromogranin A (CgA) and 24-hour urine test for 5-hydroxyindole-acetic-acid (5HIAA)
* Disease is metastatic or has recurred following surgery
* Have a CT scan performed (for the later measurement of disease volume by the core lab) within 90 days of the administration of study drug without any interventions between CT and iobenguane I 131 imaging.

All patients in Arm P and Arm C must also meet each of the following inclusion criteria:

* Provide written informed consent and are willing to comply with protocol requirements
* Are at least 18 years of age
* If female, then not of childbearing potential as documented by history (e.g., tubal ligation or hysterectomy) or is post menopausal with a minimum 1 year without menses
* If female of childbearing potential, has a negative serum HCG pregnancy test within 24 hours prior to receiving iobenguane I 131
* If female of childbearing potential, agrees to use an acceptable form of birth control, defined as abstinence or use of IUD, oral contraceptive, barrier and spermicide, or hormonal implant, throughout the study period

Exclusion Criteria:

* • Females who are nursing

  * Documented history of significant allergy that required medical intervention to shellfish, X-ray contrast media , iodine/iodides, or iobenguane
  * Administered a radioisotope within 5 effective half-lives of that radioisotope prior to study enrollment
  * Karnofsky performance status is < 60
  * Serum creatinine > 2.0 mg/dL
  * Total bilirubin > 1.5 times the upper limit of normal
  * AST/SGOT or ALT/SGPT > 3 times the upper limit of normal
  * Has received an investigational compound and/or medical device within 30 days before admission into this study
  * Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post dose follow-up examinations
  * Is determined by the Investigator that the patient is clinically unsuitable for the study
  * Has received a medication which inhibits uptake of iobenguane I 131 within 2 weeks prior to the administration of study drug. Patients must not have taken tricyclic antidepressants or related drugs within 6 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
whole body imaging immediately post-dose
whole body imaging 1 hour post-dose
whole body imaging 3 hours post-dose
whole body imaging 6 hours post-dose
whole body imaging 24 hours post-dose
whole body imaging 48 hours post-dose
whole body imaging 120 hours post-dose

SECONDARY OUTCOMES:
blood and urine samples pre-dose
blood and urine samples immediately post-dose
blood and urine samples 1 hour post-dose
blood and urine samples 3 hours post-dose
blood and urine samples 6 hours post-dose
blood and urine samples 24 hours post-dose
blood and urine samples 48 hours post-dose
blood and urine samples 120 hours post-dose
continuous urine samples at intervals of 0-6 hours, 6-24 hours, 24-48 hours, 48-72 hours, 72-96 hours and 96-120 hours post-dose
monitoring for adverse events starting when the patient consents to be in the study until 2 weeks post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ralph E Coleman, MD, Principal Investigator — Duke University